CLINICAL TRIAL: NCT04141020
Title: Effect of Sirolimus on Molecular Alterations in Cerebral Aneurysms
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Robert Starke, Assistant Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 20190857; 1R01NS111119-01A1 (NIH)
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Microsurgical Clipping Treated with Sirolimus (Experimental): Participants undergoing standard of care microsurgical clipping of unruptured cerebral aneurysm will be treated with 2 mg Sirolimus daily for 14-18 consecutive days prior to surgery.
  Interventions: Procedure: Microsurgical clipping; Drug: Sirolimus
- Endovascular Treatment Treated with Sirolimus (Experimental): Participants undergoing standard of care endovascular treatment of unruptured cerebral aneurysm procedure will be treated with 2 mg Sirolimus daily for 14-18 consecutive days prior to procedure.
  Interventions: Procedure: Endovascular treatment; Drug: Sirolimus

INTERVENTIONS:
Procedure: Microsurgical clipping — Standard of care microsurgical clipping of an unruptured cerebral artery aneurysm.
  Arms: Microsurgical Clipping Treated with Sirolimus
Procedure: Endovascular treatment — Standard of care endovascular treatment of an unruptured cerebral artery aneurysm.
  Arms: Endovascular Treatment Treated with Sirolimus
Drug: Sirolimus — Daily oral Sirolimus 2 mg tablets, adjusted as necessary per treating physician.
  Other Names: Rapamune

SUMMARY:
The objective of this study is to explore the effects of Sirolimus on the underlying molecular alterations of cerebral aneurysms.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing one of the following procedures at Jackson Memorial Hospital:

   * Clipping of an unruptured cerebral artery aneurysm
   * Endovascular treatment of unruptured cerebral aneurysms (including those receiving coiling)
2. ≥ 18 years of age
3. Willing and able to give informed consent

Exclusion Criteria:

1) Subjects meeting any of the following criteria will be excluded:

* Dissecting, traumatic, or mycotic brain aneurysm.
* Women who are pregnant, or have a positive urine or blood (β-hCG) pregnancy test.
* Women who are breastfeeding.
* Any clinically significant psychiatric or psychological disease, which would preclude the patient from completing the protocol.
* Patients with known Human Immunodeficiency Virus (HIV) infection or other known immunodeficiency.
* Patient with renal or liver failure
* Interstitial pneumonitis
* History of lymphoma
* History of skin cancer
* Hypersensitivity to sirolimus
* Severe or unstable concomitant condition disease or chronic condition, which in the opinion of the investigator could affect assessment of the safety or efficacy of study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in gene expression from control arteries. | Day 18
  Change in gene expressions will be reported as fold change from control arteries: superficial temporal artery from the same patient and the intracerebral temporal lobe artery from a different patient. Genes to be evaluated are endothelial cell marker genes such as Cluster of Differentiation (CD) 34, CD31, Von Willebrand Factor (vWF), E-selectin, Vascular Endothelial (VE)-cadherin and Endothelial Nitric Oxide Synthase (eNOS) and pro-inflammatory-matrix remodeling proliferation genes such as Matrix Metallopeptidase (MMP)3 and MMP9, Vascular Cell Adhesion Molecule (VCAM)-1, Intercellular Adhesion Molecule (ICAM), Inducible Nitric Oxide Synthase (iNOS), Membrane Cofactor Protein (MCP) and Interleukin (IL)-1ß.
Change in gene expression between blood samples. | Day 18
  Change in gene expressions will be reported as fold change of intra-aneurysmal blood to peripheral blood from the same patient. Genes to be evaluated are endothelial cell marker genes (CD34, CD31, vWF, E-selectin, VE-cadherin, and eNOS) and pro-inflammatory-matrix remodeling proliferation genes (MMP3, MMP9, VCAM-1, ICAM, iNOS, MCP, and IL-1ß).
Change in gene expression. | Day 18
  Fold change of IL-2 expression and expression of endothelial cell marker genes (CD34, CD31, vWF, E-selectin, VE-cadherin, and eNOS) and pro-inflammatory-matrix remodeling proliferation genes (MMP3, MMP9, VCAM-1, ICAM, iNOS, MCP, and IL-1ß) will be evaluated between sirolimus treated to non-treated patients.

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Starke, M.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No